CLINICAL TRIAL: NCT03652857
Title: the Effectiveness and Safety Study on Apatinib Combined With Vinorelbine Used for Driver Gene Mutation Negative Third-line and Third-line Post Progression Advanced Non-small Cell Lung Cancer
Brief Title: Apatinib Combined With Vinorelbine for Non-driver Gene Mutation Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yongchang Zhang (Other)
Responsible Party: Sponsor-Investigator, Yongchang Zhang, Professor, Hunan Province Tumor Hospital
Organization: Hunan Province Tumor Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICTOR
Record Dates: First submitted 2018-08-23; First posted 2018-08-29 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Advanced Non Small Cell Lung Cancer
Keywords: Apatinib plus Vinorelbine; NSCLC
MeSH Terms: interventions — Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib Combined With Vinorelbine (Experimental): Apatinib Combined With Vinorelbine Used for Driver Gene Mutation Negative Third-line and Third-line Post Progression Advanced Non-small Cell Lung Cancer
  Interventions: Drug: Apatinib Combined With Vinorelbine

INTERVENTIONS:
Drug: Apatinib Combined With Vinorelbine — Vinorelbine 60mg/m2 d1qweek , Apatinib 500mg po Qd,evaluate every 2months

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of Apatinib Combined With Vinorelbine Used for Driver Gene Mutation Negative Third-line and Third-line Posterior Advanced Non-small Cell Lung Cancer

DETAILED DESCRIPTION:
This efficacy and safety research plan to explore the use of Apatinib combined with Vinorelbine to driven gene mutation negative three line and three line later non-small cell lung cancer.According to the result of TAX317,the investigators expect the effective rate is 20% and 80% of degree of assurance.Single arm bilateral experiment's sample size is calculated 27, according to 10% censoring,the expected sample size is 30.

ELIGIBILITY:
Inclusion Criteria:

* 18，Pathologically proven non small cell lung cancer

  * Adenocarcinoma，No-drive gene mutaion (EGFR、ALK、ROS1） by NGS
  * Squamous cell carcinoma，no gene detection
  * Progress after second line
  * PS score >2

Exclusion Criteria:

* Patients received apatinib or Vinorelbine treatment before
* EGFR, ALK or ROS1 mutation
* Patients with contraindication of chemotherapy
* Pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
ORR | Approximately 1 years
  To measure the patients's overall response rate

SECONDARY OUTCOMES:
PFS | Approximately 1 years
  Progression free survival
OS | Approximately 1 years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Nong Yang, MD, Principal Investigator — Hunan Province Tumor Hospital
Locations (1):
- Hunan Provincal Tumor Hospital, Changsha, Hunan, China

REFERENCES:
- [Derived] Zhang X, Xiong Y, Xia Q, Wu F, Liu L, Zhou Y, Zeng L, Zhou C, Xia C, Jiang W, Liao D, Xiao L, Liu L, Yang H, Guan R, Li K, Wang J, Lei G, Zhang Y, Yang N. Efficacy and Safety of Apatinib Plus Vinorelbine in Patients With Wild-Type Advanced Non-Small Cell Lung Cancer After Second-Line Treatment Failure: A Nonrandomized Clinical Trial. JAMA Netw Open. 2020 Mar 2;3(3):e201226. doi: 10.1001/jamanetworkopen.2020.1226. PMID 32191330